CLINICAL TRIAL: NCT00839046
Title: A Community Based Participatory Research Intervention for Childhood Asthma Using Air Filters and Air Conditioners
Brief Title: A Community-based Participatory Research (CBPR) Intervention for Childhood Asthma Using Air Filters and Air Conditioners
Acronym: CAAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Toby Lewis, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01ES014566 (NIH); R01ES014566 (NIH)
Record Dates: First submitted 2009-02-05; First posted 2009-02-09 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Childhood Asthma
Keywords: Pediatric Asthma; Air Filters; Indoor Particulate Matter
MeSH Terms: interventions — Community Health Workers; Air Filters

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 Community Health Worker Intervention (Active Comparator): This is the active control group, which all 150 participants will receive. It consists of visits from trained community health workers, who will provide asthma education, as well as provision of equipment and supplies to reduce indoor environmental exposures for asthma. These will include: vacuum cleaners, mattress and pillow covers, cleaning supplies.
  Interventions: Behavioral: Community Health Worker Intervention
- 2 Air Filter (Experimental): The 50 families in the Air Filter Arm will receive an air filter in addition to the standard community health worker intervention. The Air Filter will be installed right after baseline measurements in the home.
  Interventions: Other: Air Filter
- 3 Air Filter and Air Conditioner (Experimental): Fifty families will be assigned to the "Air Filter and Air Conditioner" Arm. In addition to the standard community health worker intervention, they will receive an air filter and an air conditioner (for the warmer months).
  Interventions: Other: Air Filter and Air Conditioner

INTERVENTIONS:
Behavioral: Community Health Worker Intervention — The Community Health Worker (CHW) intervention consists of visits by CHWS to help families reduce children's exposure to common asthma triggers (allergens and irritants) in the indoor environment. The content of the CHW visits and the materials distributed will follow NHLBI Expert Panel Report 2 recommendations. Each household will receive 6 visits over a 12-month period in which the CHW will provide education on environmental triggers (e.g., reduction of dust mites, cockroaches, cat and dog dander, and environmental tobacco smoke); materials including vacuum cleaners with HEPA filters, mattress and pillow covers, and cleaning supplies; social support to the caregivers; and, if indicated, referrals to other services.
  Other Names: community health workers
  Arms: 1 Community Health Worker Intervention
Other: Air Filter — Fifty households will receive an Air Filter, in addition to receiving the standard community health worker intervention. These households will receive a HEPA room AF (Whirlpool 510 or equivalent), a relatively high capacity unit that can be quietly operated. Similar to other studies the filter will be placed in the room where the child sleeps. The HEPA AF will be installed at the beginning of the intervention period.
  Arms: 2 Air Filter
Other: Air Filter and Air Conditioner — Fifty households will receive the air filter and the air conditioner, in addition to receiving the standard community health worker intervention. The air filter will be installed at the beginning of the intervention, after baseline measurement. In the spring of the year (2009), a small window AC unit (Whirlpool Designer Style ACQ058MM or equivalent) will also be installed in the room where the child sleeps.
  Other Names: Air Conditioner; Air Filter
  Arms: 3 Air Filter and Air Conditioner

SUMMARY:
The burden of childhood asthma is borne disproportionately by children living in poverty and in urban centers, many of whom are from communities of color and are at greater risk for environmental exposures. Given the complex interaction of physical and social environmental factors on childhood asthma, there have been increasing calls for comprehensive efforts using a community-based participatory research (CBPR) approach. Community Action Against Asthma is a long standing CBPR partnership in Detroit, Michigan, composed of representatives from community-based organizations, health and human service agencies, and academia. All members of the partnership have been actively involved in the development of the CBPR project proposed here. The specific aims are: 1) to test the efficacy of air filters (AFs) separately and when combined with air conditioners (ACs) to reduce exposure to particulate matter (PM), over and above a standard community health worker home visit (standard) intervention; 2) to test the association between any reduction in PM exposure through the use of AFs separately and when combined with ACs over and above a standard intervention and health outcomes in children with asthma; 3) to elucidate the causal pathways by which any intervention-related improvements in children's asthma-related health status is occurring. One hundred and fifty households in Detroit, Michigan with at least one child with mild persistent or moderate to severe persistent asthma will be enrolled to participate in the study. Households will be randomly assigned to one of three groups: a standard household intervention (or control) group; an AF only intervention group; or an AF+AC intervention group. Extensive health and exposure measures will be undertaken during the course of the 12 -month intervention. Given the role of PM in children's asthma-related health and the higher concentrations of PM in microenvironments, there is a need to test the efficacy and efficiency of novel approaches to reducing indoor air pollutants. Doing so using a CBPR approach will enhance the relevance and ultimately the success of this proposed research.

DETAILED DESCRIPTION:
For the proposed study we will conduct a randomized controlled trial (RCT) comparing a standard community health worker home visit intervention (the standard intervention) to an Air Filter(AF) only intervention that adds the use of an AF in the child's bedroom to the standard intervention (AF only intervention) and an Air Filter(AF)+ Air Conditioner (AC) intervention that adds the use of an AF and AC in the child's bedroom to the standard intervention (AF+AC intervention) (Figure 1). We will test whether the addition of AFs (and, in the warmer months, ACs) to the standard intervention, as compared to the standard intervention will: (1) further lower children's exposure to PM (Specific Aims 1a, 1b), and (2) further improve asthma-related health status of children (Aims 2a, 2b). One hundred and fifty Detroit households with at least one child aged 6 to 12 with symptoms consistent with persistent asthma (mild, moderate, or severe) will be enrolled in the study . Following collection of baseline data, households will be randomly assigned to receive one of three interventions: the standard household intervention, the AF only intervention, or the AF+AC intervention. Participants assigned to the AF only intervention group will receive AFs at the start of the 12-month intervention (Summer/Fall 2008). Those assigned to the AF+AC intervention group will receive AFs at the start of the intervention period but ACs will not be in place during the first summer of the intervention, but will be installed in June 2009 prior to the second summer of the intervention (Figure 2). Data will be collected across all seasons (Fall 2008 through Winter 2009) which will enable us to evaluate directly the exposure and health outcome effects (Specific Aims 1a and 2a, respectively) of the addition of AFs alone to the standard intervention as well as the exposure and health outcome effects of the AFs augmented by ACs (Aims 1b, 2b). This design will also allow for comparisons, adjusted for any changes in the exposure and health status of the intervention groups, of the combined effect of the AC and AF to that of the AF alone.

ELIGIBILITY:
Inclusion Criteria:

* Residents of EastSide or Southwest Detroit
* child in the family between age of 6-12 with responses to the screening questionnaire consistent with known or probable persistent (mild, moderate, or severe) asthma

Exclusion Criteria

* the family participated in our previous intervention study in Detroit
* the family experiences continuous homelessness during the period of enrollment;
* the child spends fewer than 80% of nights at the primary household during the school year
* the child has a physical or mental handicap that would preclude successful completion of the child survey and spirometry.
* the child spends fewer than 28 consecutive nights (4 weeks) during the summer (i.e., June, July, and August) at the primary household
* the family is monolingual in a language other than English or Spanish;
* the electrical wiring of the house is inadequate for use of the air filter/air conditioner (AF/AC)
* the home lacks a closable door to the room where the child usually sleeps
* there is already an existent window AC unit in the room where the child usually sleeps
* the window in the room where the child usually sleeps will not support the addition of a window AC unit.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2007-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Improved Lung Function in Children with Asthma | End of one year of intervention

SECONDARY OUTCOMES:
Reduced Particulate Matter (PM) in the home of the children with asthma | End of one year intervention

CONTACTS AND LOCATIONS:
Overall Officials: Toby C Lewis, MD, Principal Investigator — University of Michigan School of Public Health
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States